CLINICAL TRIAL: NCT07349186
Title: Oscillometric Versus Intraarterial Blood Pressure Monitoring to Reduce Intraoperative Hypotension During Robot-Assisted Prostatectomy: A Non-Inferiority Randomized Trial
Brief Title: Oscillometric Versus Intraarterial Blood Pressure Monitoring During Robot-Assisted Prostatectomy
Acronym: PROST-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Alina Bergholz, Principal Investigator, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-101598-BOff
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillometric blood pressure monitoring (Experimental): Intraoperative blood pressure will be managed based on oscillometric blood pressure monitoring.
  Interventions: Other: Oscillometric blood pressure monitoring
- Intraarterial blood pressure monitoring (Active Comparator): Intraoperative blood pressure will be managed based on intraarterial blood pressure monitoring.
  Interventions: Other: Intraarterial blood pressure monitoring

INTERVENTIONS:
Other: Oscillometric blood pressure monitoring — In patients assigned to oscillometric blood pressure monitoring, clinicians will be blinded to intraarterial blood pressure monitoring and intraoperative blood pressure will be managed based on oscillometric blood pressure monitoring at 2.5-minute intervals.
  Arms: Oscillometric blood pressure monitoring
Other: Intraarterial blood pressure monitoring — In patients assigned to intraarterial blood pressure monitoring, intraoperative blood pressure will be managed based on intraarterial blood pressure monitoring per institutional routine.
  Arms: Intraarterial blood pressure monitoring

SUMMARY:
The PROST-BP trial is a prospective, single-center, randomized, patient-blinded, non-inferiority trial investigating whether intermittent oscillometric blood pressure monitoring is non-inferior to continuous intraarterial blood pressure monitoring in reducing intraoperative hypotension in patients having robot-assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* male patient ≥18 years
* scheduled for elective robot-assisted (Da Vinci) radical prostatectomy in steep Trendelenburg position
* planned intraarterial blood pressure monitoring

Exclusion Criteria:

* patients in whom the attending anesthesiologist considers intraarterial blood pressure monitoring to be mandatory for clinical reasons
* patients participating in another interventional trial likely to influence intraoperative blood pressure management

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average MAP <65 mmHg | From the start of surgery until the end of surgery
  Time-weighted average MAP <65 mmHg [mmHg], calculated from the start of surgery until the end of surgery (continuous endpoint)

SECONDARY OUTCOMES:
Area under a MAP <65 mmHg | From the start of surgery until the end of surgery
  Area under a MAP <65 mmHg [mmHg min] (continuous endpoint)
Total duration of MAP <65 mmHg | From the start of surgery until the end of surgery
  Total duration of MAP <65 mmHg [min] (continuous endpoint)
Number of discrete hypotensive episodes | From the start of surgery until the end of surgery
  Number of discrete hypotensive episodes, defined as MAP <65 mmHg sustained for >1 min (count endpoint)
Area above a MAP >100 mmHg | From the start of surgery until the end of surgery
  Area above a MAP >100 mmHg [mmHg min] (continuous endpoint)
Time-weighted average MAP >100 mmHg | From the start of surgery until the end of surgery
  Time-weighted average MAP >100 mmHg [mmHg], calculated from randomization until the end of surgery (continuous endpoint)
Average norepinephrine infusion rate | From the start of surgery until the end of surgery
  Average norepinephrine infusion rate [μg kg-1 min-1] (continuous endpoint)
Total volume of administered crystalloids | From the start of surgery until the end of surgery
  Total volume of administered crystalloids [ml] (continuous endpoint)

OTHER OUTCOMES:
Incidence of a composite binary outcome defined as the occurrence of at least one of the following: renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, or death | Within the first 30 postoperative days
  Incidence of a composite binary outcome defined as the occurrence of at least one of the following within the first 30 postoperative days: renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, or death (binary endpoint)
Incidence of need for renal replacement therapy | Within the first 30 postoperative days
  Incidence of need for renal replacement therapy within the first 30 postoperative days (binary endpoint)
Incidence of myocardial infarction | Within the first 30 postoperative days
  Incidence of myocardial infarction within the first 30 postoperative days (binary endpoint)
Incidence of non-fatal cardiac arrest | Within the first 30 postoperative days
  Incidence of non-fatal cardiac arrest within the first 30 postoperative days (binary endpoint)
Incidence of death | Within the first 30 postoperative days
  Incidence of death within the first 30 postoperative days (binary endpoint)
Incidence of postoperative acute kidney injury | Within the first 7 postoperative days
  Incidence of postoperative acute kidney injury within the first 7 postoperative days (binary endpoint)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany